CLINICAL TRIAL: NCT02526927
Title: Monocentric Study Evaluating Bone Microarchitecture by High Resolution Quantitative Computerized Tomography (HR-pQCT) in Young Adults and Adolescents Who Developed Anorexia Nervosa (AN) in Peri or Prepubertal Period.
Brief Title: Bone Microarchitecture Evaluation by HR-pQCT in Youngs Who Developed AN in Peri or Prepubertal Period.
Acronym: AMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1408082; 2015-A00100-49 (Other: ANSM)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; microarchitecture; prepubertal
MeSH Terms: conditions — Anorexia Nervosa | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients 20 - 30 years-old (Experimental): HR-pQCT and DEXA for measure bone quality and quantity
  Interventions: Device: HR-pQCT; Device: DEXA
- Patients 10 - 20 years-old (Experimental): Blood samples, HR-pQCT and DEXA for measure bone quality and quantity
  Interventions: Device: HR-pQCT; Device: DEXA; Other: Blood samples

INTERVENTIONS:
Device: HR-pQCT — The Xtrem CT scanco device is a HR-pQCT used for 3D bone measurements at the tibia and the radius levels in human
  Other Names: Xtrem CT scanco
Device: DEXA — The Lunar DEXA (Dual Energy X-ray Absorptiometry) is a third generation multi-captor DEXA device that allows short duration measurements (< 15 min). It measures Bone Mineral Density at the spine (L1-L4) and the femoral neck
Other: Blood samples
  Arms: Patients 10 - 20 years-old

SUMMARY:
The occurrence of anorexia nervosa (AN) during childhood or adolescence rapidly induces starvation, stop of growth and impaired mineralization of bone tissue together with an interruption of pubertal development. These consequences are initially reversible following food intake return but can lead to a more irreversible status with low height, osteoporosis and high fracture risk. The onset of the disease more and more early in life, with the first stages of puberty suggest that these consequences will be even more severe as bone resistance will be damaged by more profound effects on bone growth as well. It is therefore critical to evaluate these bone metabolism alterations in order to better manage these patients.

At every age and in every clinical circumstance either physiologic or pathologic, high resolution peripheral quantitative computerized tomography (HRpQCT) provides an evaluation of bone microarchitecture that is more informative than the global quantitative assessment given by conventional Dual Energy X-ray Absorptiometry) DEXA, with a better estimate of clinical fracture risk.

Here, we propose to measure cortical parameters, such as cortical thickness which plays a key role in bone biomechanical strength in young adults aged between 20 and 30 years-old, who had developed AN as early as the during the first stages of puberty but no longer present, compared to age-and sex-matched healthy volunteers. Other micro-architectural parameters will also be studied. In an exploratory phase, we will evaluate these bone microarchitectural parameters together with bone biological turnover markers and markers of sexual maturation in adolescents or young adults 20 years-old or less, undernourished and currently managed for AN.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years old:

  * Age > 20 and < 30 years old
  * Patients managed for AN in the pediatric or endocrinology of the university hospital of St-Etienne
  * Patients who developed AN as early as the during the first stages of puberty defined by Tanner stage 1 to 4, with a diagnosis of AN based on DSM-IV current criteria:
  * Weight loss : deny of maintaining body weight over minimal normal threshold (85 % age and height matched)
  * Intense fear of gaining weight or becoming obese despite weight insufficiency;
  * Impaired perception of weight or dysmorphophobia;
  * Excessive role of weight or body shape in self-esteem or deny of current leanness;
  * Secondary amenorrhea during 3 or more menstrual cycles in young girls or primary amenorrhea
  * Duration of AN of at least 6 months
  * BMI >85% of theoretical BMI (efficient renutrition)
* Patients less than 20 years old :

  * Age > 10 and < 20 years old
  * Patients managed for AN in the pediatric or endocrinology of the university hospital of St-Etienne
  * Patients who developed AN as early as the during the first stages of puberty defined by Tanner stage 1 to 4, with a diagnosis of AN based on DSM-IV current criteria:
  * Weight loss : deny of maintaining body weight over minimal normal threshold (85 % age and height matched)
  * Intense fear of gaining weight or becoming obese despite weight insufficiency;
  * Impaired perception of weight or dysmorphophobia;
  * Excessive role of weight or body shape in self-esteem or deny of current leanness;
  * Secondary amenorrhea during 3 or more menstrual cycles in young girls or primary amenorrhea
  * Duration of AN of at least 6 months

Exclusion Criteria:

* Renal insufficiency
* Cushing
* Dysthyroidism
* Inflammatory disease
* Pregnancy
* Lack of consent
* Subject under legal protection

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Cortical thickness | Day 1
  Cortical thickness (in mm) is a composite outcome measured with HR pQCTon 3D images of distal radius and distal tibia.

SECONDARY OUTCOMES:
Number of patients with bone degradation | Day 1
  Bone degradation is a composite outcome measured by cortical and architectural parameters measured with HR pQCTon 3D images of distal radius and distal tibia. The parameters are : Total volumetric bone mineral density (mg/ccm HA), Trabecular volumetric bone mineral density (mg/ccm HA), Cortical volumetric bone mineral density (mg/ccm HA), Number of bone trabeculae (1/mm), Trabecular thickness (mm) Cortical thickness (mm), Trabecular spacing (mm), Trabecular distribution (mm)
number of patients with osteoporosis | Day 1
  Osteoporosis is measured with DEXA. DEXA measure the Bone Mineral Density (g/cm2)
Clinical and biological phenotype of AN patients 20 years-old or less | Day 1
  Clinical and biological phenotype of AN patients 20 years-old or less is a composite factor : Pubertal stage at disease onset, Duration of AN, Height shortening compared to optimal genetically defined height, Serum levels of FGF23, Serum levels of IGF 1, Serum levels of sexual steroids (FSH, LH, oestradiol, testosterone, SeBG, AMH, inhibin B), Serum levels of bone formation and resorption markers (cross laps, osteocalcin, total alkaline phosphatases), Serum levels of leptin, Bone mineral density measured by DXA

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THOMAS, MD PhD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France